CLINICAL TRIAL: NCT00567385
Title: An Open, Multi-centre Trial Evaluating Acceptance of the New Liquid Growth Hormone Formulation - Norditropin® SimpleXx® in Children With GH Deficiency
Brief Title: Liquid Somatropin Formulation in Children With Growth Hormone Deficiency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GHLIQUID-1515
Record Dates: First submitted 2007-11-30; First posted 2007-12-04 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Growth Hormone Disorder; Growth Hormone Deficiency in Children
MeSH Terms: interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: somatropin

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to evaluate the acceptance of the new liquid growth hormone formulation, somatropin, in children with growth hormone deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Growth failure due to growth hormone insufficiency (GHD)
* Turner syndrome: established diagnosis according to sex chromosome analysis, or
* Growth retardation in children with chronic renal disorders

Exclusion Criteria:

* Pregnancy
* Breast feeding women
* Suspected or know allergy to trial product
* Participating in any other trial involving other investigational products within the last 3 months
* Previous participation in the trial
* Other daily injection therapy (non-growth hormone, e.g insulin-therapy)

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 176 (Actual)
Dates: Start 2003-03-10 (Actual); Primary Completion 2004-03-22 (Actual); Study Completion 2004-03-22 (Actual)

PRIMARY OUTCOMES:
Assessment of acceptance | after 12 weeks of treatment

SECONDARY OUTCOMES:
Safety
Adverse Events (AE)
Compliance

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Altunizade-Istanbul, Turkey (Türkiye)

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com